CLINICAL TRIAL: NCT04756453
Title: The Effect of Clip-traction on ESD Resection Time. A Randomized Controlled Trial
Brief Title: The Effect of Clip-traction on ESD Resection Time.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Richard Marsk, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-06741
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Adenoma Colon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (No Intervention): Standard endoscopic submucosal dissection
- Interventional (Active Comparator): Mandatory use of the clip-traction device
  Interventions: Device: clip-traction

INTERVENTIONS:
Device: clip-traction — A endoscopic clip with a loop of tied dental floss will be attached to the lesion. The loop will then be caught by another endoscopic clip and attached to adjacent bowel wall, thus creating tension in the tissue, making dissection easier.
  Arms: Interventional

SUMMARY:
Patients scheduled for an endoscopic submucosal dissection(ESD) in the colorectum will be randomized to the use of a traction device(consisting of an endoscopic clip with a loop of dental floss secured in the lesion to be removed, another clip will anchor the loop to adjacent bowel wall) or a standard ESD.

DETAILED DESCRIPTION:
Patients with an adenoma or an early colorectal cancer treatable with endoscopic submucosal dissection will be randomized to the use of a traction device or a standard ESD. Location, morphology and size of the lesion will be recorded. Time of the procedure will be measured using a stopwatch

ELIGIBILITY:
Inclusion Criteria:

* a lesion in the colon or rectum suitable for removal by the ESD technique

Exclusion Criteria:

* dementia
* inability to understand the written study information

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Resection speed (mm2/min) | Within completion of procedure
  Measured as area of the removed lesion divided by procedure time.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Marsk, MD,PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Endoskopicentrum Danderyds Sjukhus, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No